CLINICAL TRIAL: NCT03882372
Title: Nasal High Flow to Maintain the Benefits of Pulmonary Rehabilitation in Patients With Severe to Very Severe Chronic Obstructive Pulmonary Disease - A Randomized Controlled Study
Brief Title: Nasal High Flow to Maintain the Benefits of Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease Patients
Acronym: PPR-NHF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPR-NHF
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary rehabilitation; Nasal high flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Single blind randomized study.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be unaware of the patient's allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal high flow (Experimental): Following baseline assessment, patients randomized to the nasal high flow arm will be equipped with a nasal high flow device (myAIRVO2) administrated through the Optiflow nasal canula. Flow will be set at the highest flow tolerated (20-30 L/min): initially 30 L/min, progressively decrease if not tolerated. Temperature will be set between 34-37°C according to the tolerance : initially 37°C and decreased if not tolerated. Patients will be asked to use the device 8h per day.
  Patients under long-term oxygen will preserve their usual flow. The usual prescribed oxygen flow will then be titrated during nasal high flow to maintain the same baseline transcutaneous oxygen saturation as their conventional oxygen therapy (≥ 90%) to prevent any oxygen dilution effect of nasal high flow.
  Interventions: Device: Nasal high flow
- Usual care (No Intervention): Patient randomized to the control group will have no other specific intervention than their usual care.
  Patients under long-term oxygen will preserve their usual flow.

INTERVENTIONS:
Device: Nasal high flow — See arm description.
  Arms: Nasal high flow

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major cause of disability and mortality worldwide. This systemic disease progressively leads to dyspnea and exercise capacity impairment. Pulmonary rehabilitation effectively improves exercise capacity, dyspnea and quality of life in patients with COPD. However, its benefits progressively fade over time due to several factors such as the lack of regular exercise activity, dyspnea, airway secretions, hematosis impairment and acute exacerbations which can lead to hospitalization and accelerated muscle wasting.

Nasal high flow (NHF) is a support used to deliver heated and humidified high flow air (up to 60 L/min) through nasal canula providing promising physiological benefits such as positive airway pressure or upper airway carbon dioxide washout. It can be used in association with oxygen and offers the advantage to overtake the patient's inspiratory flow, providing a stable inspired fraction of oxygen. Nasal high flow has widely been studied in pediatric and adult intensive care units and seems better than conventional oxygen therapy and as effective as noninvasive ventilation with regards to mortality to treat hypoxemic acute respiratory failure.

More recently, several studies have shown that long-term nasal high flow could contribute to improve exercise capacity, dyspnea, airway secretion removal, hematosis, reduced acute exacerbations and subsequent hospitalizations in patients with COPD.

Based on these results, the primary aim of this study is to assess whether long-term nasal high flow treatment can help COPD patients to better maintain their endurance capacity following a course of pulmonary rehabilitation.

DETAILED DESCRIPTION:
Experimental design:

Patients achieving their last pulmonary rehabilitation session will be approached to participate in this study.

Eligible patients who agree to participate in the study and sign informed consent will perform two baseline visit assessments:

First visit: Incremental cardiopulmonary exercise testing. Second visit: Other baseline assessment (see outcome section), including a constant workload exercise testing at 75% of the maximal workload achieved during the incremental exercise testing.

Then, patients will then be randomized to one of the following two arms:

* Nasal high flow,
* Usual care.

After 6 months, patients will be invited to perform the same assessment as during the second baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease stage III to IV;
* With or without long-term oxygen therapy;
* Having completed a course of pulmonary rehabilitation within the last 4 weeks (at least 18 sessions).

Exclusion Criteria:

* Did not complete a course of pulmonary rehabilitation;
* Using noninvasive ventilation or constant positive airway pressure treatment;
* Tracheostomy;
* Nasal high flow intolerance;
* Pregnancy or likely to be;
* Unable to consent;
* Patients under guardianship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Endurance capacity | The endurance capacity will be assessed at baseline
  Patients will perform a constant workload exercise testing at 75% of the maximal workload achieved during the incremental cardiopulmonary exercise testing.
Endurance capacity | The endurance capacity will be assessed post-intervention (after 6months)
  Patients will perform a constant workload exercise testing at 75% of the maximal workload achieved during the incremental cardiopulmonary exercise testing.

SECONDARY OUTCOMES:
Quality of life: Saint George's Respiratory Questionnaire | The quality of life will be assessed at baseline
  Quality of life will be assessed using the Saint George's Respiratory Questionnaire. The score range from 0 (worst quality of life) to 100 (optimal quality of life).
Quality of life: Saint George's Respiratory Questionnaire | The quality of life will be assessed at post-intervention (after 6months)
  Quality of life will be assessed using the Saint George's Respiratory Questionnaire. The score range from 0 (worst quality of life) to 100 (optimal quality of life).
Quality of life: Chronic Obstructive Pulmonary Disease Assessement Test | The quality of life will be assessed at baseline and post-intervention for a total time frame of 6month
  Quality of life will be assessed using the Chronic Obstructive Pulmonary Disease Assessement Test
Quality of life: Chronic Obstructive Pulmonary Disease Assessement Test | The quality of life will be assessed post-intervention (after 6months)
  Quality of life will be assessed using the Chronic Obstructive Pulmonary Disease Assessement Test
Exacerbations | The number of exacerbations will be assessed for a total time frame of 6month
  The number of chronic obstructive pulmonary disease self reported exacerbations experienced by the participants during the 6 months period of follow-up will be assessed.
Hospitalizations | The number of hospitalizations will be assessed for a total time frame of 6month
  The number of chronic obstructive pulmonary disease related hospitalizations experienced by the participants during the 6 months period of follow-up will be assessed.
Muscle function (1) : quadriceps muscle (rectus femoris) cross-sectional area | The quadriceps muscle thickness will be assessed at baseline
  The quadriceps muscle thickness will be assessed using echographies.
Muscle function (1) : quadriceps muscle (rectus femoris) cross-sectional area | The quadriceps muscle thickness will be assessed at baseline and post-intervention for a total time frame of 6month
  The quadriceps muscle thickness will be assessed using echographies.
Muscle function (2) : bioimpedance | The overall muscle function using bioimpedance will be assessed post-intervention (after 6months)
  The overall muscle function will be assessed using bioimpedance (free fat mass minus total body water)
Exercise capacity | The distance performed during the six-minute walk test will be assessed at baseline
  Exercise capacity will be assessed using the six minutes walk test distance.
Exercise capacity | The distance performed during the six-minute walk test will be assessed post-intervention (after 6months)
  Exercise capacity will be assessed using the six minutes walk test distance.
Respiratory muscle function (1) : maximal inspiratory pressure | Maximal inspiratory pressure will be assessed at baseline
Respiratory muscle function (1) : maximal inspiratory pressure | Maximal inspiratory pressure will be assessed post-intervention (after 6months)
Respiratory muscle function (2) : maximal expiratory pressure | Maximal expiratory pressure will be assessed at baseline
Respiratory muscle function (2) : maximal expiratory pressure | Maximal expiratory pressure will be assessed post-intervention (after 6months)
Respiratory muscle function (3) : sniff test | Sniff test will be assessed at baseline
Respiratory muscle function (3) : sniff test | Sniff test will be assessed post-intervention (after 6months)
Parasternal electromyogram | Parasternal electromyogram will be assessed at baseline
  Parasternal electromyogram will be used to assess central output during maximal inspiratory and expiratory pressure measurement as during the sniff test. Moreover, parasternal electromyogram will be assessed both at rest and during nasal high flow (30L/min, 34°C).
Parasternal electromyogram | Parasternal electromyogram will be assessed post-intervention (after 6months)
  Parasternal electromyogram will be used to assess central output during maximal inspiratory and expiratory pressure measurement as during the sniff test. Moreover, parasternal electromyogram will be assessed both at rest and during nasal high flow (30L/min, 34°C).
Physical activity (1) : steps per day | Steps per day will be assessed during 14 days following inclusion
  The number of steps per day will be recorded over a course of 14 week days using an activity monitor.
Physical activity (1) : steps per day | Steps per day will be assessed during 14 days after 6months of intervention
  The number of steps per day will be recorded over a course of 14 week days using an activity monitor.
Physical activity (2) : time spent during activities superior to 3 metabolic equivalent per day | The time spent during activities superior to 3 metabolic equivalent per day will be assessed 14 days following inclusion
  The time spent during activities superior to 3 metabolic equivalent per day will be over a course of 14 week days
Physical activity (2) : time spent during activities superior to 3 metabolic equivalent per day | The time spent during activities superior to 3 metabolic equivalent per day will be assessed during 14 days after 6months of intervention
  The time spent during activities superior to 3 metabolic equivalent per day will be over a course of 14 week days
Quality of sleep (1) : Visual Analogue Scale | The quality of sleep using a Visual Analogue Scale will be assessed at baseline
  The quality of sleep will be assessed using a aVisual Analogue Scale (ranging from 0 to 10 with 10 indicating higher sleep quality).
Quality of sleep (1) : Visual Analogue Scale | The quality of sleep using a Visual Analogue Scale will be assessed post-intervention (after 6months)
  The quality of sleep will be assessed using a aVisual Analogue Scale (ranging from 0 to 10 with 10 indicating higher sleep quality).
Quality of sleep (2) : pittsburgh scale | The quality of sleep using the pittsburgh scale will be assessed at baseline
  The quality of sleep will be assessed using the pittsburgh scale which has been validated to assess sleep quality. The scale range from 0 (major sleep difficulties) to 21 (no difficulty).
Quality of sleep (2) : pittsburgh scale | The quality of sleep using the pittsburgh scale will be assessed post-intervention (after 6months)
  The quality of sleep will be assessed using the pittsburgh scale which has been validated to assess sleep quality. The scale range from 0 (major sleep difficulties) to 21 (no difficulty).
Adherence to treatment : days of utilization during the follow-up | The number of days that the nasal high flow device was used throughout the follow-up will be assessed post-intervention in the nasal high flow arm for a total time frame of 6 months
  The data will be retrieved from the nasal high flow device
Adherence to treatment : hours of utilization per day | The number of hours of utilization per day throughout the follow-up will be assessed post-intervention in the nasal high flow arm for a total time frame of 6 months
  The data will be retrieved from the nasal high flow device

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cuvelier, MD, PhD, Prof, Principal Investigator — Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France ; Pulmonary, Thoracic Oncology and Respiratory Intensive Care Department, Rouen University Hospital, Rouen, France; Jean-François Muir, MD, Prof, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France; Maxime Patout, MD, Msc, Study Chair — Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France ; Pulmonary, Thoracic Oncology and Respiratory Intensive Care Department, Rouen University Hospital, Rouen, France; Tristan Bonnevie, Msc, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France; Francis-Edouard Gravier, Msc, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France ; Pulmonary, Thoracic Oncology and Respiratory I
Locations (1):
- ADIR Association, Bois-Guillaume, France